CLINICAL TRIAL: NCT06462066
Title: Effectiveness, Appropriateness and Safety of GLUTACK-Glubran® Tiss 2 Surgical Glue (NBCA: n Butyl 2 Cyanoacrylate + OCA: 2-Octyl-Cyanoacrylate) Compared to GLUTACK-Glubran® 2 Device System for Mesh Fastening in Laparoscopic and Robotic Hernia Surgery (Inguinal and Ventral Hernia Repair by Sublay, Underlay and IPOM Mesh Fixation).
Brief Title: Effectiveness, Appropriateness and Safety of GLUTACK-Glubran Tiss 2 Surgical Glue Compared to GLUTACK-Glubran 2 Device System for Mesh Fastening in Laparoscopic and Robotic Hernia Surgery
Acronym: AGluTHeMFix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM SRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DGDMF/P/I.5.i.m.2/2019/1321
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Inguinal and Ventral Hernia Repair by Sublay, Underlay and IPOM Mesh Fixation
MeSH Terms: interventions — glubran 2

STUDY DESIGN:
Intervention Model Description: The study plan will include a baseline visit (V1), in which eligible patients will be randomly assigned in one of the two groups: Group 1 will apply GLUTACK/Glubran® Tiss 2 whereas Group 2 GLUTACK-Glubran® 2.
  Application of surgical glue will be done by the surgeons, after a previous appropriate training, carried out by principal investigator (standardization application mode). Trial parameters will be recorded by a clinical evaluator at 24 hours (V2), 7 days (V3), 14 days (V4), 90 days (V5) and 180 days (V6). The last evaluation will be performed at V6, after 6 month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glubran® Tiss (Experimental): The application of treatment will be performed by the Investigator that will be instructed for the application of Glutack/Glubran® Tiss 2 system.
  Glutack® is a user-friendly device for the atraumatic laparoscopic fixation of hernia mesh. Providing precise and consistent delivery of Glubran® Tiss 2/Glubran® 2 with every pull of the trigger, to minimize surgical complications and the potential pain associated with the use of tacks and staples.
  Interventions: Procedure: Experimental medical device
- Glubran® 2 (Active Comparator): The application of treatment will be performed by the Investigator that will be instructed for the application of Glutack/Glubran® 2 system.
  Glutack® is a user-friendly device for the atraumatic laparoscopic fixation of hernia mesh. Providing precise and consistent delivery of Glubran® Tiss 2/Glubran® 2 with every pull of the trigger, to minimize surgical complications and the potential pain associated with the use of tacks and staples.
  Interventions: Procedure: Comparator medical device

INTERVENTIONS:
Procedure: Experimental medical device — Open the blister and pour the sterile single-dose bottle onto the operating table in a sterile field. Before opening the single-dose bottle verify the state of fluidity of the glue and its transparency. Open the single dose of Gluban Tiss® 2. Insert the transfer tip on the single dose, grabbing it near the neck to apply adequate pressure that allows the insertion of the tip. Gradually fill the cartridge by carefully pressing on the body of the single dose.
  Other Names: Glubran Tiss
  Arms: Glubran® Tiss
Procedure: Comparator medical device — Open the blister and pour the sterile single-dose bottle onto the operating table in a sterile field. Before opening the single-dose bottle verify the state of fluidity of the glue and its transparency. Open the single dose of Glubran® 2. Insert the transfer tip on the single dose, grabbing it near the neck to apply adequate pressure that allows the insertion of the tip. Gradually fill the cartridge by carefully pressing on the body of the single dose.
  Other Names: Glubran 2
  Arms: Glubran® 2

SUMMARY:
This pre-market, prospective, randomized, non-inferiority clinical study was designed to evaluate the safety and performance/effectiveness of Glutack-Glubran® Tiss 2 system compared to Glutack-Glubran® used for mesh fixation in laparoscopic and robotic hernia surgery to obtain the indication and upgrade the medical device Glubran® Tiss 2 to class IIb.Cyanoacrylate is the generic name of a group of fast-acting adhesives such as ethyl-2-cyanoacrylate, n-butyl cyanoacrylate, 2-octy1 cyanoacrylate sold under various trade names and blend. Cyanoacrylate is a liquid acrylate monomer that polymerizes exothermically in the presence of water, especially with hydroxide ions, joining the bonded surfaces in 4-5 s and reaching the final stage in 60-90 s . It bonds body tissue excellently and shows bacteriostatic effects . The film of glue is eliminated by hydrolytic breakdown, a process whose duration varies according to tissue type and quantity .

In contrast to most cyanoacrylate glues used only for external applications as skin wound closure, Glubran® 2 is a modified n-butyl-cyanoacrylate (Glubran® 2 - N-Butyl 2 Cyanoaciylate [NBCA]+ Methacryloxysulfolane [MS]), class III medical device, CE-certified for both external and internal use .

Glubran® 2 effectiveness in repairing hernias with less post-operative pain, less complications, less hernia recurrences and a greater cost-effectiveness is largely documented . Other cyanoacrylate-based glues are authorized to fix hernia meshes, i.e.: Histoacryl (pure NBCA; classified as class IIb medical device), Liquibond FIX8 (pure NBCA; classified as class III medical device) and Ifabond (n-hexyl-cyanoacrylate; classified as class III medical device). Others are authorized to be used for specific internal indication like Omnex (2-Octyl-CyanoAcrylate [OCA] + Butyl-Lactoyl-Cyanoacrylate), which is indicated for use in vascular reconstructions. Sometimes, abroad, also some cyanoacrylate-based glues are applied for internal uses even if not authorized .

The present prospective and randomized study was aimed at comparing the effectiveness and safety of another cyanoacrylate-based glue called Glubran® Tiss 2 (NBCA + OCA), classified as class IIa surgical medical device, CE-marked (under the European Union [EU] Directive 93/42 EEC), being already authorized for use as atraumatic fixation system: Glubran® 2. Both medical devices have previously demonstrated to be well-tolerated and safe.

Glubran® 2 and Glubran® Tiss 2 were to be applied by Glutack®, a CE-marked medical device system for glue application in the surgical field. Glutack® is the related Glubran® 2/ Glubran® Tiss 2 applicator device for laparoscopic mesh fixation procedures was fabricated to offer a precise and controlled delivery of Glubran® glues .

Glubran® Tiss 2 fulfils the requirements of EU Medical Device Regulation (MDR) 2017/745 (confirmation letter received by the relative Notified Body). The composition of Glubran® Tiss 2 is obtained by mixing two different monomers of cyanoacrylate (NBCA + OCA); this gives the product a better elasticity, while maintaining high levels of tensile strength. In fact, international scientific literature has shown that the common NBCA is the cyanoacrylate molecule with the greatest tensile strength (34.27 N), low elasticity, while OCA has a lower resistance (11.27 N) but has good elastic properties. Glubran® Tiss 2 glue has a tensile strength of 27.34 N and thanks to the presence of OCA, also excellent elasticity . Among its characteristics, this formulation has haemostatic, sealing, bacteriostatic and adhesive properties. Polymerization begins 1-2 seconds after application and completes within 60 seconds. The polymerization reaction generates a temperature of approximately 45°C, which is lower than that of pure cyanoacrylates .

Glubran® Tiss 2, indicated also for use in paediatrics, is a sterile, ready for use, blended cyanacrylate adhesive to be used on the skin and mucosal tissues, which is approved as class IIa medical device, effective even in patients anticoagulated and with congenital coagulopathies .

DETAILED DESCRIPTION:
This was a pre-market, prospective, randomized, non-inferiority, clinical study aimed at evaluating the safety and performance/effectiveness of Glutack-Glubran® Tiss 2 system compared to Glutack-Glubran® 2 applied for mesh fastening in laparoscopic and robotic hernia surgery to get the indication and upgrade Glubran® Tiss 2 to class IIb. The study was conducted in seven centres in Italy and was to enroll 100 patients. Patients were to be followed for 6 months. The global duration of the trial was approximately 32 months.

According to the CIP, 6 Visits were planned over the perioperative/post operative period for each patient (after 24 hours,7, 14, 90, and 180 days).

At Visit 1 (V1, day 0, Baseline visit), patients were requested to sign the written informed consent before any procedure was performed. Patients were screened for eligibility for the study ascertaining that all inclusion criteria and no exclusion criteria were met. At V1, the Investigator recorded demographic and medical history, basal clinical assessment data and performed full physical examination and evaluation of clinical signs/symptoms.

Patients were randomly assigned (1:1 allocation ratio) to one of the two treatment groups: Glutack-Glubran® system (Group 1) or Glutack-Glubran® Tiss 2 (Group 2). The application of Glutack-Glubran® system or Glutack-Glubran® Tiss 2 was performed by the investigator, after a previous appropriate training on how to assemble/use each device.

Technical success of glue fastening was evaluated intra-operatively, the investigator registered whether mesh fixation system achieved technical success or not. Technical success was to be defined as successful hernia repair as intended, but actually defined in the present analysis as a surgical procedure with no complications within the first 24 hours after surgery and a surgeon's rating for Efficacy and Control greater than or equal to 4.At specific intervals, at V2 (24 hours), V3 (7 days), V4 (14 days), V5 (90 days) and V6 (180 days), patients were requested to return to the centre for the clinical assessments of safety, quality of life and effectiveness. As regards effectiveness, at each Visit, the area of the mesh implant was evaluated for recurrence through a specific abdominal clinical examination. In case of any suspicion of recurrence, an ultrasound or MRI was to be performed according to hospital practice to distinguish true hernia recurrences from bulging. At V6 cost effectiveness was also to be evaluated.The primary objective of the study was to assess the effectiveness of Glutack-Glubran® Tiss 2 mesh fastening in comparison with mesh fixation by Glutack-Glubran® 2 evaluated in terms of hernia recurrence rate after surgery and technical success of glue fastening (evaluated intra-operatively).

The secondary objectives were aimed at investigating the following:

1. Safety in terms of side effects
2. Cost effectiveness in terms of direct costs of intervention, operating and hospitalization times, times of return to normal activity
3. The adequacy of Glutack® medical device for the application of surgical glue for fixing the prosthesis (mesh) in terms of ease of use and satisfaction of the surgeon.

This study enrolled 107 adult patients submitted to surgical treatment for laparoceles (incisional hernia) or monolateral or bilateral inguinal hernia.

6.3.1 Inclusion Criteria

Patients could be enrolled in the investigation if they met all the following inclusion criteria:

1. No significant cardiopulmonary, hepatic, or renal impairment, and no contraindications for surgery;
2. Clinical diagnosis of:

   1. bilateral inguinal hernia eligible for minimally invasive repair (TAPP-TEP VLS/ROB)
   2. recurrent monoliteral inguinal hernia (TAPP-TEP VLS/ROB)
   3. large inguinoscrotal hernias (TAPP-TEP ROB)
   4. primary ventral hernia with defects size ≤ 7cm (IPOM-TARUP-COSTA-THT-MILOS-eMILOS VLS/ROB)
   5. primary abdominal border hernia (idem VLS/ROB)
   6. post-incisional hernia with defect size ≤ 7cm (idem VLS)
   7. post-incisional hernia and complex abdomen (RIVES-RIVES+TAR ROB)
   8. Swiss-cheese defects multiple small defects if treatable with only one mesh; if the total width of the defect is ≤ 5cm will be repaired by IPOM VLSM; if it is > 5cm will be repaired by RIVES-RIVES+TAR ROB;
3. Age > 18 years, male and Female;
4. Obese patient (BMI>35);
5. Patients with ASA grade from I to III;
6. Patients must sign and date the informed consent form prior to treatment. 6.3.2 Exclusion Criteria

Patients could not be enrolled in the investigation if they met any of the following exclusion criteria:

1. Incarcerated hernia;
2. Allergy to multiple classes of drugs, recent allergic disease, or use of drugs that are known harmful to vital organs during the 4 weeks before surgery;
3. Patients with ASA IV or V;
4. Participations in other clinical studies in the 3 months before surgery;
5. Atopic allergy history;
6. Mental illness history;
7. Diseases that may significantly increase Intra-Abdominal Pressure (IAP) and cannot be effectively controlled such as severe ascites, severe asthma caused by bronchitis, pulmonary emphysema, or urine retention caused by significant Benign Prostatic Hyperplasia (BPH);
8. Infection located at the surgical site or bacteraemia;
9. Patients with collagenopathies;
10. Relevant other concurrent diseases;
11. Patient with neurological disorders and/or mood disorders;
12. Hyperemotional patients;
13. Pregnant women.

ELIGIBILITY:
Inclusion criteria:

1. No significant cardiopulmonary, hepatic, or renal impairment, and no contraindications for surgery;
2. Clinical diagnosis of:

   1. bilateral inguinal hernia eligible for minimally invasive repair (TAPP-TEP VLS/ROB)
   2. recurrent monoliteral inguinal hernia (TAPP-TEP VLS/ROB)
   3. large inguinoscrotal hernias (TAPP-TEP ROB)
   4. primary ventral hernia with defects size ≤ 7cm (IPOM-TARUP-COSTA-THT-MILOS-eMILOS VLS/ROB)
   5. primary abdominal border hernia (idem VLS/ROB)
   6. post-incisional hernia with defect size ≤ 7cm (idem VLS)
   7. post-incisional hernia and complex abdomen (RIVES-RIVES+TAR ROB)
   8. swiss-cheese defects multiple small defects if treatable with only one mesh; if the total width of the defect is ≤ 5cm will be repaired by IPOM VLSM; if it is > 5cm will be repaired by RIVES-RIVES+TAR ROB;
3. Age > 18 years, male and female;
4. Obese patient (BMI>35);
5. Patients with ASA grade from I to III;
6. Patients must sign and date the informed consent form prior to treatment.

Exclusion criteria:

1. Incarcerated hernia;
2. Allergy to multiple classes of drugs, recent allergic disease, or use of drugs that are known harmful to vital organs during the 4 weeks before surgery;
3. Patients with ASA IV or V;
4. Participations in other clinical studies in the 3 months before surgery;
5. Atopic allergy history;
6. Mental illness history;
7. Diseases that may significantly increase Intra-Abdominal Pressure (IAP) and cannot be effectively controlled such as severe ascites, severe asthma caused by bronchitis, pulmonary emphysema, or urine retention caused by significant Benign Prostatic Hyperplasia (BPH);
8. Infection located at the surgical site or bacteraemia;
9. Patients with collagenopathies;
10. Relevant other concurrent diseases;
11. Patient with neurological disorders and/or mood disorders;
12. Hyperemotional patients;
13. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Verification of hernia recurrence at 1 day, 1 or 2 weeks, 3 months, 6 months
  A clinical examination will be conducted to evaluate recurrence. If there will be any suspicion of recurrence, an ultrasound, MRI or CT is performed according to hospital practice to distinguish true hernia recurrences from bulging. Technical success of glue fastening will be evaluated intra-operatively, the investigator will register whether mesh fixation system achieved technical success or not. Technical success is defined as successful hernia repair as intended.

SECONDARY OUTCOMES:
Clinical Safety: | Verification of Clinical safety at 1 day, 1 or 2 weeks, 3 months, 6 months
  Percentage assessment of adverse effects and events like postoperative complications including wound infection, local hematoma formation, seroma, pain, chronic pain.
Chronic pain | Verification of chronic pain at 3 months, 6 months
  Chronic pain, will be defined as moderate or greater pain in the inguinal area 3 months after surgery in which the VAS pain score was ≥4. For the evaluation of pain, an analogical visual scale will be used, identical both for the pre-operative period and for subsequent monitoring timetable. VAS pain score will be determined based on a scale of 0-10 with 0 equal to no pain and 10 equal to the worse pain imaginable.
Quality of the life | Verification of QoL at 1 day, 1 or 2 weeks, 3 months, 6 months
  Assessed by the EuraHS-QoL score. It is a method to measure the quality of life for patients before (preoperative) and after (post=operative) an operation of an abdominal wall hernia with or without an implantation of a mesh to repair the defect. It is a questionnaire developed by the Working Group of the European Registry for Abdominal Wall Hernias (EuraHS). The EuraHS-QoL score is based on a Numerical Rating Scale for three dimensions:
  1. pain at the site of the hernia or the hernia repair;
  2. restriction of activities;
  3. cosmetic discomfort;
Cost effectiveness | Verification of cost effectiveness at 1 day, 1 or 2 weeks, 3 months, 6 months
  Operating time, postoperative duration of stay, hospital costs, times to ambulatory visits, re-hospitalization for severe complications, Period to return to normal activity, measured in term of number of days after the index-procedure at which the patient resumes normal activities.
Appropriateness | Verification of Appropriateness at Intervention day during the procedure
  Appropriateness of the glue fixation system for prosthetic fixing (mesh) GLUTACK-Glubran® Tiss 2 and Glubran® assessed by the technical success of fixing the product, evaluated intra-operatively. The investigator will record if the glue fixation system for fixing the prosthesis (mesh) GLUTACK has achieved technical success or not. "Proper Use" is defined as the successful completion of all the following five steps:
  1. Attaching the cannula to handle properly;
  2. Positioning correctly the GLUTACK® device for procedure as per the user manual's instructions;
  3. Using the device's control button correctly for suitable application;
  4. Placing the cannula tip correctly at the surgical opening;
  5. Using the device for up to but not exceeding 60 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Misericordia - U.O.C Chirurgia Generale e Mini-Invasiva., Grosseto, Italy